CLINICAL TRIAL: NCT06061081
Title: A Randomized, Double-Blind (Sponsor-Unblinded), Placebo-Controlled, Adaptive Study to Investigate the Antiviral Effect, Safety, Tolerability and Pharmacokinetics of VH3739937 in Treatment-Naïve Adults Living With HIV-1
Brief Title: A Study to Investigate the Antiviral Effect, Safety, Tolerability and Pharmacokinetics of VH3739937 in in Treatment-Naive Adults Living With HIV-1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 212580; 2023-505780-37-00 (Other: European Medicines Agency)
Record Dates: First submitted 2023-09-22; First posted 2023-09-29 (Actual); Results first posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-09

CONDITIONS: HIV Infections
Keywords: VH3739937; Treatment Naïve; HIV-1
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- VH3739937 Low Dose Group (Experimental): Participants received a low dose of VH3739937 as loading Dose 1 (LD1) on Day 1, followed by a once-daily (QD) dose of VH3739937 as maintenance Dose 1 (MD1) from Days 2 through 7, where MD1 was lower than LD1. On Day 8, all participants transitioned to standard-of-care (SOC) combination antiretroviral therapy (cART) and continued study assessments through Day 25.
  Interventions: Drug: VH3739937
- VH3739937 Medium Dose Group (Experimental): Participants received a medium dose of VH3739937 as loading Dose 2 (LD2) on Day 1, followed by a QD dose of VH3739937 as maintenance Dose 2 (MD2) from Days 2 through 7, where MD2 was lower than LD2. On Day 8, all participants transitioned to SOC cART and continued study assessments through Day 25.
  Interventions: Drug: VH3739937
- VH3739937 High Dose Group (Experimental): Participants received a single high dose (Dose 3) of VH3739937 on Day 1. On Day 8, all participants transitioned to SOC cART and continued study assessments through Day 25.
  Interventions: Drug: VH3739937
- Placebo once daily (QD) (Placebo Comparator): Participants received Placebo QD from Day 1 through Day 7. On Day 8, all participants transitioned to SOC cART and continued study assessments through Day 25.
  Interventions: Drug: Placebo
- Placebo single dose (SD) (Placebo Comparator): Participants received Placebo SD on Day 1. On Day 8, all participants transitioned to SOC cART and continued study assessments through Day 25.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VH3739937 — VH3739937 will be administered.
  Arms: VH3739937 High Dose Group; VH3739937 Low Dose Group; VH3739937 Medium Dose Group
Drug: Placebo — Placebo will be administered.
  Arms: Placebo once daily (QD); Placebo single dose (SD)

SUMMARY:
The primary purpose of this study is to assess the antiviral activity of VH3739937 in Human Immunodeficiency Virus Type-1 (HIV-1) infected treatment naive (TN) participants during monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy (other than HIV infection) as determined by the Investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring
* Positive HIV antibody test
* Treatment-naïve: No Antiretrovirals (ARVs) (in combination or monotherapy) received after the diagnosis of HIV-1 infection
* Body weight ≥50.0 kilogram (kg) (110 pounds [lbs]) for men and ≥45.0 kg (99 lbs) for women and BMI for all participants within the range 18.5-35.0 kilogram per meter square (kg/m^2).
* Capable of giving signed informed consent
* Participant must be willing and able to start Combination Antiretrovial Therapy (cART) as selected with the Investigator on Study Day 8 (except in the case of early termination, clinically relevant AE/SAE, lab abnormality, the withdrawal of consent, lost to follow-up, etc., where circumstances could dictate otherwise).

Exclusion Criteria:

* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Participants with primary HIV infection, evidenced by acute retroviral syndrome (e.g., fever, malaise, fatigue, etc) and/or evidence of recent (within 3 months) documented viremia without antibody production and/or evidence of recent (within 3 months) documented seroconversion
* Myocardial infarction, acute coronary syndrome, unstable angina, stroke, transient ischemic attack, or intermittent claudication in the past 3 months
* The participant has received an investigational HIV vaccine (immunotherapeutic or immunomodulatory)
* Regular use of drugs of abuse
* Sensitivity to heparin or heparin-induced thrombocytopenia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-12-21 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2024-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (17):
- United States (3):
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Dallas, Texas
- Argentina (2):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Rosario
- GSK Investigational Site, Athens, Greece
- Italy (4):
  - GSK Investigational Site, Brescia
  - GSK Investigational Site, Genova
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Roma
- GSK Investigational Site, Warsaw, Poland
- Spain (6):
  - GSK Investigational Site, A Coruña
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Jerez de la Frontera
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Vitoria-Gasteiz

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was terminated due to Sponsor decision.
Period: Overall Study
Arm/Group | VH3739937 Low Dose Group | VH3739937 Medium Dose Group | VH3739937 High Dose Group | Placebo Once Daily (QD) | Placebo Single Dose (SD)
Started | 7 | 6 | 6 | 1 | 1
Completed | 6 | 6 | 6 | 1 | 1
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VH3739937 Low Dose Group | VH3739937 Medium Dose Group | VH3739937 High Dose Group | Placebo Once Daily (QD) | Placebo Single Dose (SD) | Total
Number analyzed (Participants) | 7 | 6 | 6 | 1 | 1 | 21
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.1 (5.52) | 38.2 (9.68) | 35.7 (14.32) | 48.0 (NA) — Standard deviation could not be calculated for a single participant. | 19.0 (NA) — Standard deviation could not be calculated for a single participant. | 34.3 (10.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 7 | 6 | 6 | 1 | 1 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 7 | 5 | 4 | 1 | 1 | 18
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 1 | 0 | 0 | 1
  Unknown | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Change From Baseline in Plasma Human Immunodeficiency Virus-1 (HIV-1) Ribonucleic Acid (RNA).
Description: Plasma samples were collected for the quantitative analysis of plasma HIV-1 RNA. The maximum change from baseline was calculated by determining the largest change from baseline value across all assessment timepoints. This is identified by subtracting the lowest post-dose visit value up to Day 8 (inclusive) from the baseline value. The baseline was defined as the most recent pre-dose assessment with a valid, non-missing value, including measurements from any unscheduled visits.
Time Frame: From Day 1 to Day 8
Population: The analysis was performed on the full analysis set (FAS) which included all randomized participants who received at least one full dose of study treatment. Only participants with data available at the specified timepoints were included in this analysis.
Measure: Mean (Standard Deviation); unit: copies/milliliter (c/mL)
Arm/Group | VH3739937 Low Dose Group | VH3739937 Medium Dose Group | VH3739937 High Dose Group | Placebo Once Daily (QD) | Placebo Single Dose (SD)
Number analyzed (Participants) | 7 | 6 | 6 | 1 | 1
copies/milliliter (c/mL) | -116909.43 (187489.611) | -130461.67 (106486.489) | -126026.67 (190725.475) | -428000.00 (NA) — Standard deviation could not be calculated for a single participant. | -14200.00 (NA) — Standard deviation could not be calculated for a single participant.

2. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) During Study Intervention Period
Description: An SAE is defined as any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant, results in abnormal pregnancy outcomes or any other situation based on appropriate medical or scientific judgement.
Time Frame: From Day 1 to Day 8
Population: The analysis was performed on the safety set which included all randomized participants who took at least 1 partial or full dose of study treatment. Only participants with data available at the specified timepoints were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | VH3739937 Low Dose Group | VH3739937 Medium Dose Group | VH3739937 High Dose Group | Placebo Once Daily (QD) | Placebo Single Dose (SD)
Number analyzed (Participants) | 7 | 6 | 6 | 1 | 1
Participants | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Reported Deaths
Time Frame: From Day 1 to Day 8
Population: The analysis was performed on the safety set. Only participants with data available at the specified timepoints were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | VH3739937 Low Dose Group | VH3739937 Medium Dose Group | VH3739937 High Dose Group | Placebo Once Daily (QD) | Placebo Single Dose (SD)
Number analyzed (Participants) | 7 | 6 | 6 | 1 | 1
Participants | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Adverse Events (AEs) Leading to Discontinuation
Description: An AE is any untoward medical occurrence (an unfavourable/unintended sign - including an abnormal laboratory finding), symptom, or disease (new or exacerbated) in a clinical study participant that is temporally associated with the study intervention. The AE may or may not be considered related to the study intervention. A participant is considered to have discontinued from the study if no new study procedure has been performed or no new information has been collected for him/her since the date of last contact.
Time Frame: From Day 1 to Day 8
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | VH3739937 Low Dose Group | VH3739937 Medium Dose Group | VH3739937 High Dose Group | Placebo Once Daily (QD) | Placebo Single Dose (SD)
Number analyzed (Participants) | 7 | 6 | 6 | 1 | 1
Participants | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of VH3739937 on QD Dosing
Description: Blood samples were collected at indicated timepoints for PK analysis.
Time Frame: Pre-dose, 1 hour (h), 2 h, 4h, 5h, 6h, 7h, 8h, 9h, 10h, 12h post-dose on Day 1
Population: The analysis was performed on the Pharmacokinetic (PK) set which included all participants in the Safety analysis set who had at least 1 PK assessment. Only participants with data available at the mentioned timepoints were included in this analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | VH3739937 Low Dose Group | VH3739937 Medium Dose Group
Number analyzed (Participants) | 7 | 6
nanogram per milliliter (ng/mL) | 397.62 (28.42) | 1225.91 (34.36)

6. Secondary Outcome: Time to Maximum Concentration (Tmax) of VH3739937 on QD Dosing
Description: Blood samples were collected at indicated timepoints for PK analysis. Tmax is defined as the time to reach maximum observed plasma concentration (Cmax).
Time Frame: Pre-dose, 1 hour (h), 2 h, 4h, 5h, 6h, 7h, 8h, 9h, 10h, 12h post-dose on Day 1
Population: The analysis was performed on the PK set. Only participants with data available at the mentioned timepoints were included in this analysis.
Measure: Median (Full Range); unit: hour (h)
Arm/Group | VH3739937 Low Dose Group | VH3739937 Medium Dose Group
Number analyzed (Participants) | 7 | 6
hour (h) | 6.00 [4.0 to 10.0] | 7.56 [4.9 to 10.1]

7. Secondary Outcome: Concentration at 24 Hours (C24) Post Dose of VH3739937 on QD Dosing
Description: C24 is defined as concentration at nominal time of 24 hours after dosing. Blood samples were collected at indicated timepoints for PK analysis.
Time Frame: At 24h post-dose on Day 1
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | VH3739937 Low Dose Group | VH3739937 Medium Dose Group
Number analyzed (Participants) | 7 | 6
ng/mL | 276.29 (102.761) | 860.17 (321.210)

8. Secondary Outcome: Area Under the Concentration-time Curve From Zero to 24h (AUC[0-24]) of VH3739937 on QD Dosing.
Description: Blood samples were collected at indicated timepoints for PK analysis.
Time Frame: Pre-dose, 1 hour (h), 2 h, 4h, 5h, 6h, 7h, 8h, 9h, 10h, 12h, 24h post-dose on Day 1
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour nanogram per milliliter (h*ng/mL)
Arm/Group | VH3739937 Low Dose Group | VH3739937 Medium Dose Group
Number analyzed (Participants) | 7 | 6
Hour nanogram per milliliter (h*ng/mL) | 6573.08 (27.55) | 20679.28 (36.73)

9. Secondary Outcome: Cmax of VH3739937 at Steady State (Cmax, ss) on QD Dosing
Description: Blood samples were collected at indicated timepoints for PK analysis.
Time Frame: Pre-dose, 1 hour (h), 2 h, 4h, 5h, 6h, 7h, 8h, 9h, 10h, 12h post-dose on Day 7
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | VH3739937 Low Dose Group | VH3739937 Medium Dose Group
Number analyzed (Participants) | 6 | 6
ng/mL | 327.09 (10.31) | 1221.20 (27.79)

10. Secondary Outcome: Tmax of VH3739937 at Steady State (Tmax, ss) on QD Dosing
Description: Blood samples were collected at indicated timepoints for PK analysis. Tmax is defined as the time to reach the maximum observed plasma concentration (Cmax).
Time Frame: Pre-dose, 1 hour (h), 2 h, 4h, 5h, 6h, 7h, 8h, 9h, 10h, 12h post-dose on Day 7
Population: as for outcome 6
Measure: Median (Full Range); unit: hour (h)
Arm/Group | VH3739937 Low Dose Group | VH3739937 Medium Dose Group
Number analyzed (Participants) | 6 | 6
hour (h) | 5.07 [2.0 to 8.0] | 7.48 [5.0 to 10.1]

11. Secondary Outcome: C24 of VH3739937 at Steady State (C24, ss) on QD Dosing
Description: Blood samples were collected at indicated timepoints for PK analysis.
Time Frame: At 24h post-dose on Day 7
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | VH3739937 Low Dose Group | VH3739937 Medium Dose Group
Number analyzed (Participants) | 6 | 6
ng/mL | 263.67 (26.493) | 937.50 (344.099)

12. Secondary Outcome: AUC(0-24) of VH3739937 at Steady State (AUC[0-24], ss) on QD Dosing
Description: Blood samples were collected at indicated timepoints for PK analysis.
Time Frame: Pre-dose, 1 hour (h), 2 h, 4h, 5h, 6h, 7h, 8h, 9h, 10h, 12h, 24h post-dose on Day 7
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | VH3739937 Low Dose Group | VH3739937 Medium Dose Group
Number analyzed (Participants) | 6 | 6
h*ng/mL | 6610.59 (16.57) | 23871.02 (30.24)

13. Secondary Outcome: Cmax Post Single Dose of VH3739937
Description: Blood samples were collected at indicated timepoints for PK analysis.
Time Frame: Pre-dose, 1 hour (h), 2 h, 4h, 5h, 6h, 7h, 8h, 9h, 10h, 12h, 24h, 48h, 72h, 96h, 120h, 144h, 168h post-dose (single dose administered on Day 1)
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | VH3739937 High Dose Group
Number analyzed (Participants) | 6
ng/mL | 2058.35 (35.50)

14. Secondary Outcome: Tmax Post Single Dose of VH3739937
Description: Blood samples were collected at indicated timepoints for PK analysis.
Time Frame: as for outcome 13
Population: as for outcome 6
Measure: Median (Full Range); unit: hour (h)
Arm/Group | VH3739937 High Dose Group
Number analyzed (Participants) | 6
hour (h) | 8.08 [6.0 to 12.0]

15. Secondary Outcome: Concentration at 168 Hours (C168) Post Single Dose of VH3739937
Description: C168 is defined as concentration of VH3739937 at a nominal time of 168 hours after dosing. Blood samples were collected at indicated timepoints for PK analysis.
Time Frame: At 168 hours post-dose (single dose administered on Day 1)
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | VH3739937 High Dose Group
Number analyzed (Participants) | 6
ng/mL | 297.25 (35.19)

16. Secondary Outcome: Area Under the Concentration-time Curve From Zero to 168h [AUC(0-168)] Post Single Dose of VH3739937
Description: Blood samples were collected at indicated timepoints for analysis.
Time Frame: as for outcome 13
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | VH3739937 High Dose Group
Number analyzed (Participants) | 6
h*ng/mL | 144443.90 (39.51)

ADVERSE EVENTS:
Time Frame: AEs were reported from Day 1 to Day 25. SAEs and All-cause mortality were reported from the signing of the informed consent form (a period starting up to 14 days before the first dose on Day 1) to Day 25.
Description: SAEs and AEs were reported for the Safety set. Safety set included all randomized participants who took at least 1 partial or full dose of study treatment.
Arm/Group | VH3739937 Low Dose Group | VH3739937 Medium Dose Group | VH3739937 High Dose Group | Placebo Once Daily (QD) | Placebo Single Dose (SD)
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6 | 0/6 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/7 | 1/6 | 0/6 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 3/7 | 2/6 | 5/6 | 0/1 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VH3739937 Low Dose Group (N=7) | VH3739937 Medium Dose Group (N=6) | VH3739937 High Dose Group (N=6) | Placebo Once Daily (QD) (N=1) | Placebo Single Dose (SD) (N=1)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VH3739937 Low Dose Group (N=7) | VH3739937 Medium Dose Group (N=6) | VH3739937 High Dose Group (N=6) | Placebo Once Daily (QD) (N=1) | Placebo Single Dose (SD) (N=1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Energy increased (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gonococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-10-06): https://cdn.clinicaltrials.gov/large-docs/81/NCT06061081/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-30): https://cdn.clinicaltrials.gov/large-docs/81/NCT06061081/SAP_001.pdf